CLINICAL TRIAL: NCT01341574
Title: Influence of Prism Adaptation on Spatial Neglect in the Early Versus Delayed Phase After Stroke: a Randomized, Placebo-controlled Trial
Brief Title: Early Versus Delayed Treatment of Unilateral Neglect After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Fund for Scientific Research, Flanders, Belgium (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011/161; G.0906.10 (Other Grant/Funding Number: FWO)
Record Dates: First submitted 2011-04-18; First posted 2011-04-25 (Estimated); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Spatial Neglect After Stroke
Keywords: spatial neglect; stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- Early phase, experimental (Experimental): Neglect patients, randomized in the experimental group (Prism adaptation, optical shift of 10 degrees) in the early phase after stroke.
  Interventions: Procedure: Prism adaptation with optical shift of 10 degrees.
- Delayed phase, experimental (Experimental): Neglect patients, randomized in the experimental group (Prism adaptation, optical shift of 10 degrees) in the delayed phase after stroke.
  Interventions: Procedure: Prism adaptation with optical shift of 10 degrees.
- Early phase, placebo (Placebo Comparator): Neglect patients, randomized in the placebo group (Prism adaptation, optical shift of 0 degrees) in the early phase after stroke.
  Interventions: Procedure: Prism adaptation optical shift of 0 degrees.
- Delayed phase, placebo (Placebo Comparator): Neglect patients, randomized in the placebo group (Prism adaptation, optical shift of 0 degrees) in the delayed phase after stroke.
  Interventions: Procedure: Prism adaptation optical shift of 0 degrees.
- Delayed phase postural, experimental (Experimental): Neglect patients, randomized in the experimental group (Prism adaptation, optical shift of 10 degrees) in the delayed phase after stroke. In this group, postural aspects are taken into account.
  Interventions: Procedure: Prism adaptation with optical shift of 10 degrees.

INTERVENTIONS:
Procedure: Prism adaptation with optical shift of 10 degrees. — Prism adaptation with optical shift of 10 degrees.
  Arms: Delayed phase postural, experimental; Delayed phase, experimental; Early phase, experimental
Procedure: Prism adaptation optical shift of 0 degrees. — Prism adaptation with optical shift of 0 degrees.
  Arms: Delayed phase, placebo; Early phase, placebo

SUMMARY:
'Unilateral neglect' is a disorder that occurs regularly after stroke. It is caused by right- as well as left-sided brain lesions, but more often by right-sided lesions. Patients with this disorder neglect the contralesional side of space and/or their body. Their body axis is often shifted ipsilesionally. A specific disorder that can appear in neglect patients is 'contraversive pushing': a postural deviation to the neglected side because the patient pushes himself away from the ipsi- to the contralesional side.

One of the most promising neglect interventions is prism adaptation (PA): inducing an optical shift of the visual field by means of prism glasses. This results in a modulation of brain areas involved in neglect and in an improvement of the neglect symptoms and postural deviation.

Research questions:

1. Which period is best suited to maximize therapeutic effects? In this respect the effects of early and delayed PA will be compared, regarding neglect-, postural and cerebral measures.
2. Which factors lead to a less favorable treatment outcome or to therapy resistance for PA?
3. Will the impact of PA be larger if postural factors are taken into account in the prism therapy?

ELIGIBILITY:
Inclusion Criteria:

* male or female
* > 17 years of age
* stroke patients with clinical neglect, demonstrated by neglect tests

Exclusion Criteria:

* severe ocular abnormalities
* not being able to perform prism adaptation or neglect tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
effect of prism adaptation | Briefly after and 3 months after therapy cycle.
  The effect of Prism Adaptation (PA) will be evaluated regarding the degree of neglect, postural control and cerebral functioning, briefly after the therapy cycle and 3 months later. Briefly after the PA sessions and three months later, in patients in the early as well as the delayed phase after stroke:
  * early: PA starting within 4 weeks after stroke;
  * delayed: PA starting 2 months after stroke;
  * OR divided in an early and a delayed group according to the median.

SECONDARY OUTCOMES:
The degree of well-being. | Briefly after and 3 months after therapy cycle.
  Questionnaires about emotional and functional status.
  Briefly after the Prism Adaptation (PA) sessions and 3 months later, in patients in the early as well as the delayed phase after stroke:
  * early: PA starting within 4 weeks after stroke;
  * delayed: PA starting 2 months after stroke;
  * OR divided in an early and a delayed group according to the median.

CONTACTS AND LOCATIONS:
Overall Officials: Guy Vingerhoets, Ph.D., Professor, Principal Investigator — University Ghent
Locations (3):
- Belgium (3):
  - Rehabilitation Hospital "Hof ter Schelde", Antwerp
  - Ghent University Hospital, Center for Locomotor and Neurological Rehabilitation, Ghent
  - Ghent University Hospital, Department of Neurology, Ghent